CLINICAL TRIAL: NCT07093580
Title: Phase 1 Study of a Long-acting Injectable S-892216 in Healthy Adult Participants
Brief Title: Study of S-892216 Long-acting Injectable (LAI) in Healthy Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2316T1711
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Healthy Participants
Keywords: First-in-human (FIH); Long-acting injectable (LAI) formulation; S-892216; S-892216-LAI; Severe acute respiratory syndrome coronavirus 2; SARS-CoV-2 infection; Novel Coronavirus; Coronavirus Disease 2019; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Single Ascending Dose) (Experimental): Participants will receive a single dose of S-892216-LAI or placebo on Day 1.
  Interventions: Drug: S-892216-LAI; Drug: Placebo
- Part 2 (Multiple Ascending Dose) (Experimental): Participants will receive multiple doses of S-892216-LAI or placebo on Day 1 and Day 85 in treatment periods 1 and 2, respectively.
  Interventions: Drug: S-892216-LAI; Drug: Placebo

INTERVENTIONS:
Drug: S-892216-LAI — S-892216-LAI injection will be administered per schedule specified in the arm description.
Drug: Placebo — Physiological saline will be administered per schedule specified in the arm description.

SUMMARY:
The purpose of this study is to investigate the safety, tolerability, and pharmacokinetics (PK) of single- and multiple-dose administration of S-892216-LAI in healthy adults.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) ≥18.5 and ≤32.0 kilograms (kg)/square meter (m^2)

Key Exclusion Criteria:

* Presence or history of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, neurological, or ophthalmological (for example, increased intra-ocular pressure) disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data per the investigator's assessment.
* History of cancer except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Require medication or other treatment (for example, dietary restrictions or physical therapy).
* Participated in any other clinical study involving an investigational study intervention or any other type of medical research within 30 days, or 5 times the half-life of the investigational drug, before signing of the informed consent form (ICF) for this study or who are currently participating in such a study.
* Positive test results of the following at screening or within 6 months prior to administration of study intervention: hepatitis B surface antigen (HBsAg); hepatitis C virus antibody (HCV); and human immunodeficiency virus (HIV) antigen/antibody.
* Positive severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) reverse transcription polymerase chain reaction (RT-PCR) test result, positive transcription-mediated amplification test result, positive antigen test result, or any other test approved according to local regulations at check in for each period on admission.
* Known allergy/sensitivity or any hypersensitivity to components of S-892216-LAI or placebo for S-892216-LAI.
* Used cannabis (medical or recreational), tobacco, or nicotine-containing products (including e-cigarettes, pipe tobacco, cigar, chewing tobacco, nicotine patch, and nicotine gum) within 6 months prior to admission.

Note: Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2027-05-26 (Estimated); Study Completion 2027-05-26 (Estimated)

PRIMARY OUTCOMES:
Part: Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Day 1 through Day 364
Part 2: Number of Participants With TEAEs | Day 1 through Day 448

SECONDARY OUTCOMES:
Part 1: Maximum Plasma Concentration (Cmax) of S-892216 and its Metabolites | Day 1 (pre-administration, up to 12 hours post-administration) through Day 364
Part 2: Cmax of S-892216 and its Metabolites | Day 1 (pre-administration, up to 12 hours post-administration) through Day 70 in Treatment Period 1 and Day 85 (pre-administration, up to 12 hours post-administration) through Day 448 in Treatment Period 2
Part 1: Time to Reach Cmax (Tmax) of S-892216 and its Metabolites | Day 1 (pre-administration, up to 12 hours post-administration) through Day 364
Part 2: Tmax of S-892216 and its Metabolites | Day 1 (pre-administration, up to 12 hours post-administration) through Day 70 in Treatment Period 1 and Day 85 (pre-administration, up to 12 hours post-administration) through Day 448 in Treatment Period 2
Part 1: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration After Dosing (AUC0-last) of S-892216 and its Metabolites | Day 1 (pre-administration, up to 12 hours post-administration) through Day 364
Part 2: AUC0-last of S-892216 and its Metabolites | Day 1 (pre-administration, up to 12 hours post-administration) through Day 70 in Treatment Period 1 and Day 85 (pre-administration, up to 12 hours post-administration) through Day 448 in Treatment Period 2

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - ICON Clinical Research: Lenexa, Lenexa, Kansas
  - ICON Clinical Research: Salt Lake City, Salt Lake City, Utah